CLINICAL TRIAL: NCT02204969
Title: Transcranial Magnetic Stimulation (TMS) and Lithium Water for Treatment of Alzheimer Patients
Brief Title: LIWA for Treatment of Alzheimer Patients
Acronym: LIWA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Society Of Thermalism And Climatology Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 822429989
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial magnetic stimulation (Sham Comparator): All participants will receive standard medical therapy for AD. In addition, patients recruited for the study will receive 16 sessions of TMS with the H2 coil over 8 weeks. The first group will receive excitatory stimulation of 10 Hz over the prefrontal and parietal cortex, the second group will receive inhibitory stimulation of 1 Hz over similar brain areas and control patients will receive the same amount of Sham sessions. Patient will receive 3 treatments per week in the first 3 weeks and then 1 treatment per week for additional 4 weeks.
  Interventions: Device: Transcranial Magnetic stimulation
- lithia water (Placebo Comparator): * Experimental: Lithia spring water Lithia water (active) for 4 weeks then placebo water for 4 weeks Intervention: Dietary Supplement: Lithia water
  * Placebo Comparator: Natural spring water Placebo water for 4 weeks then lithia water (active) for 4 weeks Intervention: Dietary Supplement: Natural spring water with negligible lithium levels
  Interventions: Dietary Supplement: Lithia water

INTERVENTIONS:
Dietary Supplement: Lithia water — * Experimental: Lithia spring water Lithia water (active) for 4 weeks then placebo water for 4 weeks Intervention: Dietary Supplement: Lithia water
  * Placebo Comparator: Natural spring water Placebo water for 4 weeks then lithia water (active) for 4 weeks Intervention: Dietary Supplement: Natural spring water with negligible lithium levels
  Other Names: pring Mineral water
  Arms: lithia water
Device: Transcranial Magnetic stimulation — All participants will receive standard medical therapy for AD. In addition, patients recruited for the study will receive 16 sessions of TMS with the H2 coil over 8 weeks. The first group will receive excitatory stimulation of 10 Hz over the prefrontal and parietal cortex, the second group will receive inhibitory stimulation of 1 Hz over similar brain areas and control patients will receive the same amount of Sham sessions. Patient will receive 3 treatments per week in the first 3 weeks and then 1 treatment per week for additional 4 weeks.
  Other Names: novel coil design (H2)
  Arms: Transcranial magnetic stimulation

SUMMARY:
The thermal therapy combined with magnetic fields and ozone has a direct effect on patients with dementia and Alzheimer's with a regression of more than 60% of them

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the leading cause of dementia and cognitive deteriorating in the advanced age. This main target of this study is to determine the safety and efficacy of transcranial magnetic stimulation (TMS) using novel coil design (H2) for stimulation of deep brain structures concomitantly with regular treatment in Alzheimer's disease (AD) patients. TMS acts by generating magnetic fields in the brain which simulate neuro-chemical changes and stimulate neuronal activity translating into increased secretion of growth factors such as brain derived neurotropic factor (BDNF). Hence it is postulated that TMS will have a positive effect on the cognitive and behavioral symptoms of patients with AD and may ameliorated the progression of the disease. The treatment is non-invasive, with no significant side effects, and no need of hospitalization or anesthesia. The trial is phase II double blind study including 100 AD patients ages between 50 to 80 with mild or moderate AD (Mini Mental State Examination [MMSE] 16 to 26) divided into 3 groups. All participants will receive standard medical therapy for AD. In addition, patients recruited for the study will receive 16 sessions of TMS with the H2 coil over 8 weeks. The first group will receive excitatory stimulation of 10 Hz over the prefrontal and parietal cortex, the second group will receive inhibitory stimulation of 1 Hz over similar brain areas and control patients will receive the same amount of Sham sessions. Patient will receive 3 treatments per week in the first 3 weeks and then 1 treatment per week for additional 4 weeks. Patients will be evaluated before the treatments, after 8 weeks of treatment and after another 8 weeks without treatment. The evaluations will include cognitive function according to ADAS-COG and MMSE, Activity of daily living (ADL) functions according to ADSC-ADL, behavioral function according to the Neuropsychiatric Inventory (NPI), depression according to the Cornell Scale for Depression in Dementia (CSDD), care giver satisfaction according to the RUD LITE scale and computerized cognitive evaluation according to the NEXING battery. We expect that the cognitive, behavioral and ADL functions will improve better in the study group as compared to the Sham treated group. From previous trial of TMS in neurological patients, although not in AD, we anticipate that adverse events rate will be similar between groups proving the safety of deep TMS treatment in patients with AD. In case our hypothesis will be proven, deep TMS treatment will be added as an important modality to the conventional therapy of AD patients.

All patients will be received 500 mcg/d of lithium as supplement nutritional in form spring mineral water

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50-85.
2. Diagnosed with Alzheimer's disease for at least half a year (by the DSM-IV criteria).
3. Scored 16-26 on the MMSE.
4. Received drug therapy for their disease, with each treatment having been administered at an acceptable dosage for at least 5 weeks.
5. Existence of a routine therapist for changes or adverse effects reports.
6. Existence of Alzheimer diagnosis by CT or MRI tests.
7. Answered in the negative to all questions in the pre-TMS treatment safety questionnaire.
8. Gave their oral and written consent to participate in the trial.

Exclusion Criteria:

1. An additional neurological disorder.
2. Severe psychiatric disorder.
3. Uncontrolled hypertension, beyond 170/110.
4. History of epilepsy, seizure, or heat convulsion or History of epilepsy or seizure in first degree relatives.
5. History of head injury or stroke.
6. History of metal implants in the head (except dental fillings)or History of surgery entailing metallic implants or known history of any metallic particles in the eye, implanted cardiac pacemaker, cochlear implants, use of neuro stimulators, or any medical pumps.
7. History of migraines in the last six months.
8. History of drug or alcohol abuse.
9. Inadequate communication with examiner.
10. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it.
11. Inability to sign a consent form.
12. Leukemia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning score by ADAS-COG | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Garis Silega, Dr, Principal Investigator — American Society of Thermalism and Climatology
Locations (1):
- Gaviota Clinic, Newark, New Jersey, United States